CLINICAL TRIAL: NCT06035380
Title: The Effect of Aromatherapy to Women With Vasomotor Complaints on Menopausal Quality
Brief Title: The Effect of Aromatherapy to Women With Vasomotor Complaints on Menopausal Quality of Life and Vasomotor Symptoms
Acronym: Aromatherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Gülsen Müsteyde Altan, lecturer, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EasternMU-SBF-HB-GMAD-01
Record Dates: First submitted 2023-06-08; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Aromatherapy
Keywords: Aromatherapy, Vasomotor Symptoms

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rose oil (Experimental): rose oil will be used
  Interventions: Other: rose oil group
- mint oil (Experimental): mint oil will be used
  Interventions: Other: mint oil group
- plasebo (Placebo Comparator): drinking water will be used
  Interventions: Other: placebo group

INTERVENTIONS:
Other: placebo group — aromatherapy
  Arms: plasebo
Other: mint oil group — aromatherapy
  Arms: mint oil
Other: rose oil group — aromatherapy
  Arms: rose oil

SUMMARY:
Evaluation of the effect of aromatherapy applied to women with vasomotor complaints on menopausal quality of life and vasomotor symptoms.

DETAILED DESCRIPTION:
Menopause, ovarian failure due to loss of follicular function of the ovaries accompanied by estrogen deficiency, causes permanent cessation of menstruation and loss of reproductive function. The period in which irregularities in the menstrual cycle begin to appear and the chance of fertility decreases is defined as the premenopausal period. During this period, vasomotor complaints occur. vasomotor complaints; It is reported as hot flashes, sweating and night sweats . It has been reported that women experience an average of 4-5 hot flashes per day , and this number reaches 20 in some women . These changes are usually the most severe and disturbing findings two or three years before menopause and can continue in later years . Studies have reported that vasomotor complaints negatively affect women's quality of life.

Application methods of aromatherapy with many therapeutic benefits, massage oil, face cream/oil, gel, body bath, hand and foot baths, compresses, hot towels, aromatic sprays, bath salt, inhalations (direct bottle, sniffing salt, drip on handkerchief), steam inhalation, facial mist, diffusion (diffuser, nebulizer, candle), ointment, mouthwash . Studies have also reported that aromatherapy methods used during menopause reduce vasomotor complaints and positively affect quality of life .

Evaluating and supporting women in line with the holistic nursing approach is among the responsibilities of nurses. Nurses' development of appropriate care standards in line with these goals constitutes an important step for women to step into a healthy and high-quality old age. Women's health nurses should provide care, counseling and training to increase the quality of life of women who spend one-third of their life in the menopausal period .

Studies have reported that aromatherapy has a positive effect on quality of life. However, studies on this subject in Türkiye and the Turkish Republic of Northern Cyprus are quite limited.

Purpose of the research; This study will be conducted to evaluate the effect of aromatherapy applied to women with vasomotor complaints on menopausal quality of life and vasomotor symptoms.

The population of the study will consist of women living in the Turkish Republic of Northern Cyprus, Famagusta District and reporting more than 5 vasomotor complaints according to the Visual Analog Scale. The sample size was determined as 66 by G*Power analysis. Three groups will be formed by randomization method from the people who agreed to participate in the study, while rose oil will be used in the first group, peppermint oil will be used in the second group, and the third group will form the placebo group.

Essential oils to be used in groups to be treated with aromatherapy are rose and mint oils. In addition to the cooling effect of rose oil, it is known that thanks to its pleasant smell, it helps the user to feel good and is also effective in reducing menopausal symptoms. At the same time, peppermint oil is stated to revitalize the body, increase energy level, provide refreshment and reduce menopausal symptoms . It will be used after diluting by adding 10 ml of black cumin oil as carrier oil to 2 drops of rose and mint oils to be used in the study.

In 2021, the researcher completed the 90-hour theoretical and 16-hour applied aromatherapy training program, coordinated by Riccon Academy-Bern-Schweiz and Adamer training center, and received her certificate.

The placebo group will be asked to use the spray whenever they complain of hot flashes, using drinking water.

With this randomized controlled study, it is aimed to evaluate the effect of aromatherapy applied to women with vasomotor complaints on menopausal quality of life and vasomotor symptoms, and to provide evidence for the care to be offered to menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Being able to speak Turkish,
* Getting a score above 5 in VAS
* Not to be allergic to the aromatherapy oils to be applied,
* Lack of sense of smell,
* Accepting to work with essential oils to be studied,
* Not having entered menopause naturally,
* Not using hormone replacement therapy,
* Not using complementary alternative therapy,
* Women who do not have a psychiatric problem,

Exclusion Criteria:

-Wanting to leave the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — * pre menopause
  * menopause
  * post menopause
Enrollment: 66 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
VISUAL ANALOGUE SCALE (VAS) | Baseline, 1 day
  VAS is used to convert some values that cannot be measured numerically. This scale is a safe, easily applicable test that has proven itself for a very long time and has been accepted in all the world literature. The test has no language and its ease of implementation is an important advantage. It was used in this study to determine how much hot flashes complaints experienced by women affect their lives. It was explained to the women that one end of the scale did not affect their life at all (0), and that it affected their life too much as they approached the other end (10). The women were asked to mark the number on a divided line with numbers from 0 to 10, and how much they thought their hot flashes had affected their lives.
Introductory Information Form | Baseline, 1 day
  women's socio-demographic characteristics , physical characteristics , pregnancy and birth information (pregnancy). number of people living together, spousal support, menstrual pattern, last menstrual period, age of mother's menopause, chronic diseases, smoking and alcohol use, vasomotor complaints, use of CAM and nursing support are included in a total of 27 questions.
Hot Flashes Scale Specific to Menopause | Baseline, 1 day, the ninetieth day
  The Menopause-Specific Hot Flashes Scale is used to measure the effect of hot flashes on overall quality of life (item 10) and nine specific activities (item 1-item 9). Nine specific activities: work, social activities, leisure activities, sleep, mood, concentration, relationships with others, sexuality, enjoyment of life. How much hot flashes affect the woman's life during the last two weeks is evaluated by numerical rating method from 0 to 10. A value of 0 means "not at all affected" and a value of 10 means "very much affected". The total score is calculated by adding the numerical values of each item.
Menopause-Specific Quality of Life Scale | Baseline, 1 day, the ninetieth day
  It is a 29-item Likert-type scale. The scale consists of four domains: vasomotor, psychosocial, physical and sexual. Vasomotor domain (questions 1-3), Psychosocial domain (questions 4-10), Physical space (questions 11-26), Sexual domain (questions 27-29), Each sub-domain score in the scale is ranked from 1 to 8. 1 point indicates that there is no problem with that. A score of 2 indicates that the problem exists, exists, but is not bothersome at all. Scores between 3 and 8 indicate the severity of the existing problem and its increasing degrees.
Aromatherapy Form | 12 week
  The usage time and usage amount of the aromatherapy oil will be filled on the aroma therapy form for 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohebitabar S, Shirazi M, Bioos S, Rahimi R, Malekshahi F, Nejatbakhsh F. Therapeutic efficacy of rose oil: A comprehensive review of clinical evidence. Avicenna J Phytomed. 2017 May-Jun;7(3):206-213. PMID 28748167
- [Background] Johnson A, Roberts L, Elkins G. Complementary and Alternative Medicine for Menopause. J Evid Based Integr Med. 2019 Jan-Dec;24:2515690X19829380. doi: 10.1177/2515690X19829380. PMID 30868921
- [Background] Short M. Menopause, mood and management. Climacteric. 2003 Aug;6 Suppl 2:33-6. PMID 14669842